CLINICAL TRIAL: NCT01706003
Title: The Utility of Telemedicine in the Management of Migraine: A Pilot Study :MK0974-071-00
Brief Title: The Utility of Telemedicine in the Management of Migraine
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Deborah Friedman, Primary Investigator, MD, Neurology and Neurotheraputics, University of Texas Southwestern Medical Center
Other Study IDs: MK0974-071-00; MERCK (Other: MISP)
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-09

CONDITIONS: Migraine Headaches
Keywords: Migraine; Headaches; Telemedicine
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Telemedicine Group: People who suffer from Migraine Headaches who own a computer and have internet access and will be treated via telemedicine for migraine headaches
- In-Office Group: People who suffer from Migraine Headaches who own a computer and have internet access and will be treated in the clinician's office for migraine headaches

SUMMARY:
Patients will be randomly assigned to receive their follow-up care via telemedicine or in-office visits.

DETAILED DESCRIPTION:
After obtaining informed consent, patients will be randomly assigned to receive their follow-up care via telemedicine or in-office visits. All subjects will complete a MIDAS questionnaire and allodynia questionnaire at their initial visit. Follow-up visits will be scheduled at 4-6 weeks, 3, 6, 9 and 12 months. In-person follow-up visits will be conducted in the standard fashion of the current physician's practice, with the initial intake conducted by an ophthalmic technician or resident, followed by the physician visit. Telemedicine visits will be conducted by the physician and recorded. Similar information will be gathered in both groups including: current medications, interim medical and headache history (including visits to the ED or hospitalizations for headache), description of headache, response to treatment (including adverse reactions), allergies, blood pressure and weight. Subjects randomized to telemedicine will be asked to have their blood pressure and weight measured within 5 days of their telemedicine session at a location convenient to them. We will record the length of each visit. Subjects in the in-person group, will be queried about travel time, and the total amount of time for the visit, and any activities missed to attend the visit. We will also ask about other costs associated with attending the office visit, such as child care.

At the one-year follow-up visit, subjects will complete the MIDAS, allodynia questionnaire, Modified Group Health Association of America's Consumer Satisfaction scale, and have the opportunity to express their views on the aspect of care received in a semi-structured interview. The follow-up questionnaires may be completed on line (telemedicine group, optional for in-person group) or on paper (in-person group). Headache diaries will be provided on line or may be done on paper, a smartphone, or a computer program of the subject's choosing.

All subjects will be able to access the physician by telephone, using MyChart, or with additional non-study visits as needed.

Subjects will be responsible for the cost of the medications, treatments prescribed, and laboratory monitoring needed for their condition.

Support staff will be available to help set up the video system for subjects assigned to the telemedicine group who are in need of assistance.

ELIGIBILITY:
Inclusion Criteria:• Ages 18 - 89 years

* Diagnosis of migraine with or without aura, menstrual migraine, hemiplegic migraine
* Able to provide informed consent
* Able, in the opinion of the investigator, to reliably perform all aspects of the study
* Ownership of or access to a computer and high speed internet

Criteria for Exclusion of Subjects:

* Age less than 18 years
* Headache type is not migraine
* No ownership or access to a computer or high speed internet
* Unfamiliar with basic computer operations or uncomfortable using a computer
* Unwilling to participate
* Unable to read English (because of assessment tools)
* History of another medical, psychiatric, social or behavioral problem that, in the opinion of the investigator, makes it unlikely that they will be able to complete the study activities. Questions regarding mood and anxiety are asked of all patients as part of their initial evaluation for headache.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be diagnosed with Migraine Headaches
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-10; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Friedman, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Universit of Texas Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friedman DI, Rajan B, Seidmann A. A randomized trial of telemedicine for migraine management. Cephalalgia. 2019 Oct;39(12):1577-1585. doi: 10.1177/0333102419868250. Epub 2019 Aug 26. PMID 31450969

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | In-Office Group | Telemedicine Group
Started | 23 | 22
Completed | 12 | 18
Not Completed | 11 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Not scheduled | 3 | 0
Not completed — Lost to Follow-up | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-Office Group | Telemedicine Group | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 2 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45
Migraine Disability Assessment Score (MIDAS) [Mean (Full Range); unit: units on a scale] — The Migraine Disability Assessment Score (MIDAS) has a scale range of 0-270. Lower values represents a better outcome, higher values represents a worse outcome.
  units on a scale | 40.5 [3 to 161] | 65 [11 to 192] | 47.9 [3 to 192]

OUTCOME MEASURES:

1. Primary Outcome: Assess the Utility of Telemedicine for Follow-up Care in a Headache Medicine Practice
Description: Percentage of completed scheduled study visits for each group.
Time Frame: One Year
Measure: Number; unit: percentage of scheduled appointments
Arm/Group | In-Office Group | Telemedicine Group
Number analyzed (Participants) | 12 | 18
percentage of scheduled appointments | 87 | 92.7

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | In-Office Group | Telemedicine Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 3/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Office Group (N=23) | Telemedicine Group (N=22)
Hospital admission (Nervous system disorders) | 0 (0) | 3 (5) — Hospitalized for headache treatment as part of routine clinical care

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-02-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT01706003/Prot_SAP_000.pdf